CLINICAL TRIAL: NCT03738644
Title: Near-infrared Spectroscopy in Endovascular Treatment (Danish: Nær-infrarød Spektroskopi Ved endovaskulær Trombektomi)
Brief Title: Monitoring Stroke Patients With Near-infrared Spectroscopy Before, During and After Endovascular Treatment
Status: Completed | Type: Observational
Sponsor: Helle Klingenberg Iversen (Other)
Responsible Party: Sponsor-Investigator, Helle Klingenberg Iversen, Senior neurologist, Head of Stroke Unit, Associate Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-18028704; H-18028704 (Other: Scientific Ethics Committee, The Capital Region of Denmark); VD-2018-269 (I-suite: 6509) (Other: Danish Data Protection Agency)
Record Dates: First submitted 2018-10-17; First posted 2018-11-13 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Ischemic Stroke
Keywords: Endovascular treatment; Near-infrared spectroscopy; Intra-operational monitoring
MeSH Terms: conditions — Ischemic Stroke | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples, serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Monitoring with near-infrared spectroscopy — No interventions are used. Stroke patients are examined with near-infrared spectroscopy (NIRS). NIRS examinations are done with Octamon system (Artinis Medical Systems, Elst, The Netherlands) consisting of 8 transmitters emitting infrared light of 760 and 850 nm and 2 receivers measuring oxygenated and deoxygenated hemoglobin in the frontal cortex.
  Examination protocol can be found in detailed description.

SUMMARY:
The purpose of this study is to examine the hemodynamics of stroke patients with near-infrared spectroscopy before, during and after endovascular treatment and their relations to disabilities and mortality 3 months after treatment.

DETAILED DESCRIPTION:
Endovascular treatment is the revascularization after ischemic stroke due to large-artery occlusion by mechanical removal of thrombi with an intraarterial catheter. The area around the infarction called the penumbra, which has partial blood supply by collateral vessels, can thereby be salvaged and the neuronal function restored. EVT lowers the disabilities and the morbidity if it is performed within 6 hours of onset or within 24 hours in stroke patients with a significant penumbra (Rodrigues, Neves et al. 2016).

However, complications can arise during EVT including critically failing CBF, intracranial hemorrhage and embolization of the thrombus to more peripheral vessels, which can all result in further brain damage.

To avoid these repercussions or detect them as fast as possible as well as detecting successful interventions, a suitable method for monitoring CBF over time is needed. NIRS is a commonly applied method that examines CBF in the cerebral cortex, which has already been used as intraoperative monitoring during abdominal and cardiac surgery (Yu, Zhang et al. 2018), but only in minor studies of EVT patients, where results have been very promising and associated to long-term outcomes (Hametner, Stanarcevic et al. 2015, Ritzenthaler, Cho et al. 2017). NIRS exploits that absorption of infrared light is only changed by hemoglobin, which can therefore by measured over time. NIRS is a non-invasive and safe method that measures oxygenated and deoxygenated hemoglobin in the cerebral cortex (Ferrari and Quaresima 2012).

Cerebral autoregulation (CA) is a complex mechanism that maintains an relatively constant and adequate CBF, which is often impaired in acute stroke patients (Paulson, Strandgaard et al. 1990). The nature of CA can be examined with NIRS (Obrig, Neufang et al. 2000, Reinhard, Wehrle-Wieland et al. 2006, Schytz, Hansson et al. 2010, Zweifel, Dias et al. 2014) and impairment can be shown (Li, Wang et al. 2010, Han, Li et al. 2014, Han, Zhang et al. 2014, Phillip and Schytz 2014). NIRS examinations of CA has never been done during EVT and the relation between changes in CA and patient outcome remains unknown.

This leads to the following hypothesis:

* CBF and CA can be monitored with NIRS before, during and after EVT and detect complications and successful EVTs.
* CBF and CA during and after EVT can be associated to the disabilities and mortality of stroke patients 3 months after the treatment.

The investigators will examine stroke patients who receive EVT with NIRS. The equipment will be placed on participants forehead when they arrive to the department and monitored for up to 2 hours after EVT. A 20-minute follow-up NIRS examinations will be done at 24 hours and 3 months after EVT. National Institute of Health Stroke Scale (NIHSS) will be performed before and after EVT, at 24 hours and 3 months after EVT. Participants will be assessed for functioning level and scored for independence with Modified Ranking Scale and screened for new vascular events, complications related to EVT and death by cause after 3 months.

To satisfy power calculations, 100 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients receiving endovascular treatment

Exclusion Criteria:

* Premorbid mRS > 3
* Acute EEG examinations within 2 hours after EVT
* Neurosurgical evacuation within 2 hours after EVT
* Remaining life expectancy < 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who could be candidates for endovascular treatment in Region Zealand and The Capital Region of Denmark are assessed in Rigshospitalet, yearly around 200 patients. If endovascular treatment is attempted, subjects will be included. Only ischemic stroke patients with large-vessel occlusion will be eligible for endovascular treatment.
  Only patients fulfilling the inclusion criteria and not the exclusion criteria are eligible. Patients will be enrolled before consent is given. Consent is obtained after endovascular treatment after oral and written information is provided. Recruitment is approved by Ethics Committee.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Oxygenated hemoglobin ratio of total hemoglobin before, during and after endovascular treatment | From onset of examination before EVT, during EVT and up to 2 hours after EVT.
  Variability in oxygenated hemoglobin from onset of examination before EVT until end of examination up to 2 hours after EVT

OTHER OUTCOMES:
Oxygenated hemoglobin ratio of total hemoglobin before and after endovascular treatment | Baseline before EVT is initiated, last part of monitoring period (up to 2 hours) after EVT and 20 min. recordings 24 hours and 90 days after EVT.
  Changes in oxygenated hemoglobin ratio of total hemoglobin from baseline (before EVT) to last part of monitoring period (up to 2 hours) and to 20 min. recordings at 24 hours and 90 days.
Oxygenated hemoglobin before and after endovascular treatment | From onset of examination before EVT, during EVT and up to 2 hours after EVT.
  Variability in oxygenated hemoglobin from onset of examination before EVT until end of examination up to 2 hours after EVT
Oxygenated hemoglobin before and after endovascular treatment | Baseline before EVT is initiated, last part of monitoring period (up to 2 hours) after EVT and 20 min. recordings 24 hours and 90 days after EVT.
  Changes from baseline (before EVT) to last part of monitoring period (up to 2 hours) and to 20 min. recordings at 24 hours and 90 days.
Independence assessed with modified Ranking Scale (mRS) | 90 days after EVT
  mRS 90 days after EVT. The mRS scale runs from 0-6, running from perfect health without symptoms (score of 0) to death (score of 6).
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Degree of disabilities assessed by National Institute of Health Stroke Scale (NIHSS) | Changes from just before EVT to 2 hours, 24 hours and 90 days after EVT
  Changes is NIHSS from before EVT to after EVT.
  National Health Institute Stroke Scale (NIHSS): Stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.
Composite vascular outcome of new events | 90 days after EVT
  New stroke or transitory cerebral ischemia, acute coronary syndrome or operation for peripheral artery disease.
Complications related to EVT | 90 days after EVT
  Any complications related to EVT 90 days after procedure.
Mortality | 90 days after EVT
  Death by cause at 90 days after EVT

CONTACTS AND LOCATIONS:
Overall Officials: Helle K Iversen, DMSc, Principal Investigator — Department of Neurology, Rigshospitalet
Locations (1):
- Department of Neurology, Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hametner C, Stanarcevic P, Stampfl S, Rohde S, Veltkamp R, Bosel J. Noninvasive cerebral oximetry during endovascular therapy for acute ischemic stroke: an observational study. J Cereb Blood Flow Metab. 2015 Nov;35(11):1722-8. doi: 10.1038/jcbfm.2015.181. Epub 2015 Aug 5. PMID 26243709
- [Background] Ritzenthaler T, Cho TH, Mechtouff L, Ong E, Turjman F, Robinson P, Berthezene Y, Nighoghossian N. Cerebral Near-Infrared Spectroscopy: A Potential Approach for Thrombectomy Monitoring. Stroke. 2017 Dec;48(12):3390-3392. doi: 10.1161/STROKEAHA.117.019176. Epub 2017 Oct 31. PMID 29089454
- [Background] Ferrari M, Quaresima V. A brief review on the history of human functional near-infrared spectroscopy (fNIRS) development and fields of application. Neuroimage. 2012 Nov 1;63(2):921-35. doi: 10.1016/j.neuroimage.2012.03.049. Epub 2012 Mar 28. PMID 22510258
- [Background] Paulson OB, Strandgaard S, Edvinsson L. Cerebral autoregulation. Cerebrovasc Brain Metab Rev. 1990 Summer;2(2):161-92. PMID 2201348
- [Background] Obrig H, Neufang M, Wenzel R, Kohl M, Steinbrink J, Einhaupl K, Villringer A. Spontaneous low frequency oscillations of cerebral hemodynamics and metabolism in human adults. Neuroimage. 2000 Dec;12(6):623-39. doi: 10.1006/nimg.2000.0657. PMID 11112395
- [Background] Reinhard M, Wehrle-Wieland E, Grabiak D, Roth M, Guschlbauer B, Timmer J, Weiller C, Hetzel A. Oscillatory cerebral hemodynamics--the macro- vs. microvascular level. J Neurol Sci. 2006 Dec 1;250(1-2):103-9. doi: 10.1016/j.jns.2006.07.011. Epub 2006 Oct 2. PMID 17011584
- [Background] Schytz HW, Hansson A, Phillip D, Selb J, Boas DA, Iversen HK, Ashina M. Spontaneous low-frequency oscillations in cerebral vessels: applications in carotid artery disease and ischemic stroke. J Stroke Cerebrovasc Dis. 2010 Nov-Dec;19(6):465-74. doi: 10.1016/j.jstrokecerebrovasdis.2010.06.001. PMID 20864356
- [Background] Zweifel C, Dias C, Smielewski P, Czosnyka M. Continuous time-domain monitoring of cerebral autoregulation in neurocritical care. Med Eng Phys. 2014 May;36(5):638-45. doi: 10.1016/j.medengphy.2014.03.002. Epub 2014 Apr 1. PMID 24703503
- [Background] Han Q, Li Z, Gao Y, Li W, Xin Q, Tan Q, Zhang M, Zhang Y. Phase synchronization analysis of prefrontal tissue oxyhemoglobin oscillations in elderly subjects with cerebral infarction. Med Phys. 2014 Oct;41(10):102702. doi: 10.1118/1.4896113. PMID 25281981
- [Background] Han Q, Zhang M, Li W, Gao Y, Xin Q, Wang Y, Li Z. Wavelet coherence analysis of prefrontal tissue oxyhaemoglobin signals as measured using near-infrared spectroscopy in elderly subjects with cerebral infarction. Microvasc Res. 2014 Sep;95:108-15. doi: 10.1016/j.mvr.2014.08.001. Epub 2014 Aug 10. PMID 25117487
- [Background] Li Z, Wang Y, Li Y, Wang Y, Li J, Zhang L. Wavelet analysis of cerebral oxygenation signal measured by near infrared spectroscopy in subjects with cerebral infarction. Microvasc Res. 2010 Jul;80(1):142-7. doi: 10.1016/j.mvr.2010.02.004. Epub 2010 Feb 13. PMID 20156461
- [Background] Phillip, D. and H.W. Schytz, Spontaneous Low Frequency Oscillations in Acute Ischemic Stroke ? A Near Infrared Spectroscopy (NIRS) Study. Journal of Neurology & Neurophysiology, 2014. 05(06).
- [Result] Rodrigues FB, Neves JB, Caldeira D, Ferro JM, Ferreira JJ, Costa J. Endovascular treatment versus medical care alone for ischaemic stroke: systematic review and meta-analysis. BMJ. 2016 Apr 18;353:i1754. doi: 10.1136/bmj.i1754. PMID 27091337
- [Result] Yu Y, Zhang K, Zhang L, Zong H, Meng L, Han R. Cerebral near-infrared spectroscopy (NIRS) for perioperative monitoring of brain oxygenation in children and adults. Cochrane Database Syst Rev. 2018 Jan 17;1(1):CD010947. doi: 10.1002/14651858.CD010947.pub2. PMID 29341066
- [Derived] Heiberg AV, Lukassen TG, Truelsen TC, Borgwardt HG, Benndorf G, Solling C, Schytz HW, Moller K, Hansen K, Iversen HK. Dynamic cerebral autoregulation during and 3 months after endovascular treatment in large vessel occlusion stroke. Sci Rep. 2025 Aug 19;15(1):30289. doi: 10.1038/s41598-025-14672-y. PMID 40830559